CLINICAL TRIAL: NCT05599360
Title: Vyxeos for Induction of Newly Diagnosed Low- or Intermediate-risk AML Patients, Age 18-70. A Pilot Study
Brief Title: Vyxeos for Induction of Low- or Intermediate-risk.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Chezi Ganzel, Director, Hematology Day Care, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0463-20 SZMC
Record Dates: First submitted 2022-01-20; First posted 2022-10-31 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vyxeos (Experimental)
  Interventions: Drug: Vyxeos; Drug: Mylotarg

INTERVENTIONS:
Drug: Vyxeos — Vyxeos (daunorubicin and cytarabine) liposome for injection
  Other Names: cpx-351
Drug: Mylotarg — Gemtuzumab ozogamicin is an antibody-drug conjugate (ADC) composed of the CD33-directed monoclonal antibody (hP67.6; recombinant humanized immunoglobulin [Ig] G4, kappa antibody produced by mammalian cell culture in non-secreting 0 (NS0) cells) that is covalently linked to the cytotoxic agent N-acetyl gamma calicheamicin. Gemtuzumab ozogamicin consists of conjugated and unconjugated gemtuzumab. The conjugated molecules differ in the number of activated calicheamicin derivative moieties attached to gemtuzumab. The number of conjugated calicheamicin derivatives per gemtuzumab molecule ranges from predominantly zero to 6, with an average of 2 to 3 moles of calicheamicin derivative per mole of gemtuzumab.
  Other Names: gemtuzumab ozogamicin

SUMMARY:
Vyxeos Vyxeos is a liposomal-encapsulated combination of cytarabine and daunorubicin, at a molar ratio of 5:1. Delivery of the 5:1 molar ratio seems to prevent antagonistic drug-drug interactions and the liposomal encapsulation increases the plasma half-life of cytarabine and daunorubicin and leads to drug accumulation within the bone marrow (BM).

Despite previous results that highlighted the advantage of Vyxeos for sAML, it is intuitively likely that this powerful drug is also suitable for non-sAML. The mechanism of action is relevant for every AML. Following the FDA approval of the drug for sAML we would like to evaluate its efficacy for low or intermediate risk fms-like tyrosine kinase 3 (FLT3)-negative de novo AML patients. This consideration is particularly relevant by the inclusion of young AML patients in the study.

Gemtuzumab ozogamicin (GO) Gemtuzumab ozogamicin (Mylotarg) - an anti-cluster of differentiation 33 (CD33) monoclonal antibody linked to calicheamicin, was approved for the treatment of newly diagnosed AML patients, when given as a combination with the '7+3' regimen.

One of the goals of the current study is to examine the feasibility and efficacy of the combination of Mylotarg plus Vyxeos.

Minimal/ measurable residual disease (MRD) Minimal or measurable residual disease (MRD) denotes the presence of leukemia cells down to levels of 1:10-4 to 1:10-6, compared with 1:20 in morphology-based assessments. MRD can be evaluated using a variety of multiparameter flow cytometry (MFC) and molecular methods. There are no data regarding the achievement or impact of MRD using Vyxeos as induction therapy. The current trial will address this issue.

Purpose of this Trial The current study is designed to examine the response rate of the Vyxeos as induction therapy for newly diagnosed low/intermediate risk AML patients in the 'real world' setting. Patients will receive the same induction therapy that they were to receive had they not entered this study (cytarabine /daunorubicin ± Mylotarg) but the combination of cytarabine /daunorubicin will be given in the unique formulation of Vyxeos. In addition to classic CR+CRi evaluation, MFC MRD evaluation, using an centralized, internationally recognized laboratory, will be done at the end of induction. In addition, this pilot study will also provide clinical safety information about the combination of Vyxeos with Mylotarg.

DETAILED DESCRIPTION:
Introduction Induction therapy Currently, most physicians treating 'fit' patients with acute myeloid leukemia (AML) employ an anthracycline plus cytarabine ('7+3' regimen) as induction therapy. In the past few years 2 new drugs were approved as adjuncts to the '7+3' regimen for treatment of fit patients; Midostaurin- a FLT3 inhibitor and gemtuzumab ozogamicin- an anti-CD33 monoclonal antibody linked to chemotherapy. It has been postulated that using the same drugs as in the '7+3' regimen but at a fixed molar ratio of cytarabine and daunorubicin will increase the CR rate and improve minimal residual disease and disease free survival (DFS).

Vyxeos

Vyxeos is a liposomal-encapsulated combination of cytarabine and daunorubicin, at a molar ratio of 5:1. Delivery of the 5:1 molar ratio seems to prevent antagonistic drug-drug interactions and the liposomal encapsulation increases the plasma half-life of cytarabine and daunorubicin and leads to drug accumulation within the bone marrow (BM). Two randomized controlled trials have been reported in newly diagnosed AML patients:

A phase II, multicenter, randomized, open-label trial studied the efficacy and safety of Vyxeos among newly diagnosed AML patients, age 60-75. The study compared 1-2 induction courses of Vyxeos with '7+3' (daunorubicin dose of 45-60 mg/m2). Patients were allowed to receive 1-2 consolidation courses of Vyxeos (in the investigational arm) and low dose cytarabine with/without daunorubicin or intermediate dose cytarabine (in the control arm). The primary end-point was defined as response rate; complete remission (CR) + CR with incomplete hematologic recovery (CRi). 127 patients were enrolled and randomized in 2:1 ratio. The study showed an increased response rate (CR+CRi of 66.7% vs. 51.2%) in the investigational arm but without statistical significance (p=0.7). A planned sub-group analysis of secondary AML (sAML) patients revealed a more impressive, still non-significant, response rate advantage to the Vyxeos patients (57.6% vs. 31.6%, p=.06) but with significant overall survival (OS) superiority (median 12.1 vs. 6.1 months, HR = 0.46, p=.01).

The phase III trial was an open-labeled randomized trial that enrolled only sAML patients, age 60-75, with the exception of patients with antecedent myeloproliferative neoplasm. Patients received 2-3 cycles (1-2 induction courses and 1 consolidation) of either '7+3' with daunorubicin 60 mg/m2 or Vyxeos. The primary end-point was defined as OS. A total of 309 patients were enrolled and randomized in a 1:1 ratio. This study showed a significant OS (median of 9.56 vs. 5.95 months, HR=0.69, p=.005) and CR+CRi rate (47.7% vs. 33.3%, p=.016) advantage for the patients who received the Vyxeos. These results led the Food and Drug Administration (FDA), in August 2017, to approve the drug for use in the treatment of newly diagnosed therapy-related AML (tAML) and AML with myelodysplasia-related changes (MRC).

Despite the results that highlighted the advantage of Vyxeos for sAML, it is intuitively likely that this powerful drug is also suitable for non-sAML. The mechanism of action is relevant for every AML. Following the FDA approval of the drug for sAML we would like to evaluate its efficacy for low or intermediate risk FLT3-negative de novo AML patients. This consideration is particularly relevant by the inclusion of young AML patients in the study.

Gemtuzumab ozogamicin (GO) Gemtuzumab ozogamicin (Mylotarg) - an anti-CD33 monoclonal antibody linked to calicheamicin, was approved for the treatment of newly diagnosed AML patients, when given as a combination with the '7+3' regimen.

The French Alfa-0701 study evaluated the safety and efficacy of GO administered in a fractionated dosing regimen (3 mg/m² administered on Days 1, 4, and 7) when added to the standard '7+3' regimen. Patients with a CR or CR with incomplete platelet recovery (CRp) received consolidation therapy with 2 courses of treatment including daunorubicin plus cytarabine with or without GO, based on their initial randomization. The primary end point was event free survival (EFS) which was longer in the GO arm; median of 17.3 months (95% combination index (CI): 13.4-30.0) vs 9.5 months (95% CI: 8.1-12.0). 3-years EFS was achieved by 39.8% of the GO arm compared to 13.6% of the control arm. OS was better in the GO arm (27.5 vs. 21.8 months) but have not reached statistical significance (HR 0.807, 95% CI: 0.596-1.093, p=0.1646)5. A meta-analysis of GO in combination with chemotherapy for newly diagnosed AML patients concluded that GO does not increase the CR rate but decreases the relapse rate and improves the OS. The drug is ineffective in high risk patients.

One of the goals of the current study is to examine the feasibility and efficacy of the combination of Mylotarg plus Vyxeos.

Minimal/ measurable residual disease (MRD) Several factors present at diagnosis of AML, including cytogenetics, molecular genetics, and age, have been associated with prognosis. Increasing evidence now indicates that the ability to identify residual disease far below the morphology-based 5% blast threshold is an important tool for refining the approach to risk classification. Minimal or measurable residual disease (MRD) denotes the presence of leukemia cells down to levels of 1:10-4 to 1:10-6, compared with 1:20 in morphology-based assessments. MRD can be evaluated using a variety of multiparameter flow cytometry (MFC) and molecular methods. There are no data regarding the achievement or impact of MRD using Vyxeos as induction therapy. The current trial will address this issue.

Purpose of this Trial The current study is designed to examine the response rate of the Vyxeos as induction therapy for newly diagnosed low/intermediate risk AML patients in the 'real world' setting. Patients will receive the same induction therapy that they were to receive had they not entered this study (cytarabine /daunorubicin ± Mylotarg) but the combination of cytarabine /daunorubicin will be given in the unique formulation of Vyxeos. In addition to classic CR+CRi evaluation, MFC MRD evaluation, using an centralized, internationally recognized laboratory, will be done at the end of induction. In addition, this pilot study will also provide clinical safety information about the combination of Vyxeos with Mylotarg.

Gender and Ethnicity Entry to this study is open to both men and women, and to persons of any racial or ethnic group. We are aware of no data that would lead us to expect differential treatment effects by gender and ethnicity and therefore have not incorporated separate accrual goals for these subgroups.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of AML (>20% blasts in blood or BM)
2. Favorable or intermediate risk cytogenetics

Exclusion criteria:

1. Acute promyelocytic leukemia with recurring translocations involving Retinoic Acid Receptor Alpha (RARA)
2. Acute leukemias of ambiguous lineage
3. Therapy-related myeloid neoplasms
4. Background of myelodysplastic syndrome or myeloproliferative neoplasm
5. FLT3-Internal tandem duplications (ITD) mutation with any allelic ratio
6. AML with Adverse cytogenetic risk (ELN 2017)
7. Eastern Cooperative Oncology Group (ECOG) performance status 3-4
8. Previous treatment with radiation therapy or cytotoxic chemotherapy (treatment with corticosteroids or hydroxyurea will not exclude the patient)
9. Age<18 or >70
10. Serum creatinine ≥ 2.0 mg/dl or creatinine clearance < 50 ml/min within 14 days of registration
11. Direct bilirubin ≥2.0 g/dl, or alkaline phosphatase/ serum glutamic-oxaloacetic transaminase (SGOT) > 4xupper limit of normal within 14 days of registration
12. Left ventricular ejection fraction (LVEF)<45%
13. Pregnant or breastfeeding women
14. Blastic transformation of chronic myelogenous leukemia (CML)
15. Secondary AML (defined as prior chemotherapy-induced or evolved from myelodysplastic syndrome or myeloproliferative neoplasm)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2028-09-07 (Estimated); Study Completion 2028-09-07 (Estimated)

PRIMARY OUTCOMES:
Response rate for low/intermediate risk AML after induction with Vyxeos | Up to 1 month
  Complete Remission (CR) and Complete Remission with incomplete Hematologic Recovery (CRi) rate.
Safety of the combination of Vyxeos plus Mylotarg as per CTCAE v5.0. | Up to 5 years
  Number and severity of adverse events (AEs) and adverse events serious adverse events (SAEs) of participants with Vyxeos plus Mylotarg treatment. AEs and SAEs of both treatment and non-treatment-related will be collected at REDCAP project and assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
MFC MRD level after Vyxeos without Mylotarg treatment | Up to 1 month
  Multiparameter Flow Cytometry Minimal Residual Disease (MFC MRD) levels before and after Vyxeos will be collected.
MFC MRD levels after Vyxeos with Mylotarg treatment | Up to 1 month
  Multiparameter Flow Cytometry Minimal Residual Disease (MFC MRD) levels before and after Vyxeos and Mulotarg will be collected.
Disease free survival (DFS) post Vyxeos ± Mylotarg induction therapy | Up to 5 years
  Disease free survival (DFS) post Vyxeos ± Mylotarg induction therapy by testing disease status as schedule:
  During 1st year - every 3 months During 2nd year - every 6 months For the following 3 years, once a year, or in a case known of disease relapse.
Overall survival (OS) post Vyxeos ± Mylotarg induction therapy | Up to 5 years
  Overall survival (OS) post Vyxeos ± Mylotarg induction therapy by testing survival status monthly.

CONTACTS AND LOCATIONS:
Overall Officials: Chezi Ganzel, DR, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) available to other researchers.